CLINICAL TRIAL: NCT01830712
Title: A Long-Term Assessment of Physical Activity, Range of Motion, and Functional Status Following Elective Orthopedic Surgery in Hemophilia Patients With Inhibitors. A Retrospective Follow-up Assessment to F7HAEM/USA/3/USA and F7HAEM/USA/4/USA
Brief Title: A Long-term Assessment of Physical Activity, Range of Motion, and Functional Status Following Elective Orthopedic Surgery in Hemophilia Patients With Inhibitors
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: F7HAEM-3864; U1111-1114-9206 (Other: WHO)
Record Dates: First submitted 2013-04-10; First posted 2013-04-12 (Estimated); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Congenital Bleeding Disorder; Haemophilia A With Inhibitors; Haemophilia B With Inhibitors
MeSH Terms: interventions — Factor VII

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chart review
  Interventions: Drug: eptacog alfa (activated)

INTERVENTIONS:
Drug: eptacog alfa (activated) — A review of retrospectively longitudinal data gathered in the routine follow-up from a subset of patients who underwent EOS in studies F7HAEM/USA/3/USA and F7HAEM/USA/4/USA (NCT01561391). Data will be compiled, analysed, and reported in aggregate form.

SUMMARY:
This study is conducted in the United States of America (USA). The aim of this study is to assess the long-term (5+ years) postoperative functional outcomes of elective orthopaedic surgery (EOS) patients from previously reported studies F7HAEM/USA/3/USA and F7HAEM/USA/4/USA (NCT01561391) and furthermore to assess the impact of EOS on psychosocial outcomes, frequency of bleeding episodes and durability of joint surgery.

ELIGIBILITY:
Inclusion Criteria:

* Haemophilia patients with inhibitors who have had EOS during their participation in F7HAEM/USA/3/USA and F7HAEM/USA/4/USA (NCT01561391)

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Haemophilia patients with inhibitors who had EOS during their participation in F7HAEM/USA/3/USA or F7HAEM/USA/4/USA (NCT01561391).
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2011-04; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Long-term changes in general mobility/ambulation/activity | From pre-operative (baseline) functional status and up to at least 5 years

SECONDARY OUTCOMES:
Long-term changes in work/school attendance | From pre-operative (baseline) functional status and up to at least 5 years
Long-term changes in employment status | From pre-operative (baseline) functional status and up to at least 5 years
Long-term changes in body mass index (BMI) | From pre-operative (baseline) functional status and up to at least 5 years
Long-term changes in complications related to surgical procedure and/or prostheses | From pre-operative (baseline) functional status and up to at least 5 years
Overall frequency of bleeding episodes | From pre-operative (baseline) functional status and up to at least 5 years
Number of joint infections | From pre-operative (baseline) functional status and up to at least 5 years
Number of treatment types (on demand, prophylaxis) | From pre-operative (baseline) functional status and up to at least 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Clinical Trial Call Center, Princeton, New Jersey, United States

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com